CLINICAL TRIAL: NCT06825780
Title: Short Term Outcomes of Primary Percutaneous Coronary Intervention (PCI) Patients Presented with Acute Heart Failure in Assuit University Heart Hospital
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sanaa Gamal Abdel Nasser, cardiology, Assiut University
Other Study IDs: PCI.HF
Record Dates: First submitted 2025-02-08; First posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Primary Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Observational study outcome of PCI in patients presented with acute heart failure

ELIGIBILITY:
Inclusion Criteria:

* age more than 18 years
* acute heart failure
* PCI

Exclusion Criteria:

* NSTEMI
* end stage renal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: assiut university heart hospital
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-03-03 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
hospital mortality and complication post PCI | within 3 month
  number of mortality cases

SECONDARY OUTCOMES:
major adverse cardiac events | within 3 month
  myocardial infarction heart failure

CONTACTS AND LOCATIONS:
Overall Officials: doaa fouad abdelgaoad, staff, Principal Investigator — staff
Locations (1):
- Heart Hospital, Asyut, Heart Hospital, Egypt

REFERENCES:
- [Background] Lembo NJ, Karmpaliotis D, Kandzari DE. CTO PCI Procedural Planning. Interv Cardiol Clin. 2012 Jul;1(3):299-308. doi: 10.1016/j.iccl.2012.04.002. Epub 2012 Jun 5. PMID 28582014